CLINICAL TRIAL: NCT03186430
Title: A Practice-Provider-Parent-Adolescent Intervention to Increase HPV Vaccination
Brief Title: PreTeenVax Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Robert Bednarczyk, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00090382; K01AI106961 (NIH)
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Human Papilloma Virus
Keywords: Vaccine; Vaccination; Behavioral Research; Adolescent; Health Promotion; Public Health

STUDY DESIGN:
Intervention Model Description: This study uses a cluster-randomized design where six health provider practices are randomized to the intervention or control arm where all participants in the respective practices will receive the behavioral intervention or the standard information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Vaccine Promotion Package (Experimental): The pediatric practices randomized to this arm will receive the comprehensive adolescent vaccine promotion package. Practice physicians and staff will be familiarized with each component, and practices will be instructed to implement each vaccine-promotion component to the best of their ability.
  Interventions: Behavioral: Comprehensive Vaccine Promotion Package
- Standard Vaccination Promotion (No Intervention): The pediatric practices randomized to the control arm will not receive the comprehensive vaccine promotion package and will instead be instructed to continue offering their standard adolescent vaccination promotion practices to adolescent patients.

INTERVENTIONS:
Behavioral: Comprehensive Vaccine Promotion Package — Practice-level components: Periodic feedback on adolescent immunization coverage. Assistance with implementing and utilizing standing orders for adolescent vaccine administration in the practice, utilizing standardized materials as provided by the Centers for Disease Control and Prevention and the Immunization Action Coalition. Identification of an immunization champion to facilitate immunization activities in the practice. Linkage to peer-to-peer training on adolescent vaccination through the Georgia Educating Providers In their Communities (EPIC) program.
  Provider-level components: Providers will receive standardized talking points, vaccine promotion scripts and answers to frequently asked questions, with training on how best to discuss, recommend and answer questions about vaccines.
  Patient/Parent-level components: An iPad tablet-based educational presentation will be provided for parents while they are waiting with their adolescent child in the examination room.
  Arms: Comprehensive Vaccine Promotion Package

SUMMARY:
The primary research aim of this project is to test the effectiveness of a comprehensive, evidence-based vaccine promotion toolkit implemented in the pediatric healthcare setting on increasing the likelihood that adolescents in Georgia will initiate and complete the Human Papillomavirus (HPV) vaccine series. Secondary research aims include assessing the impact of the comprehensive toolkit on 1) patient and parent knowledge and attitudes regarding HPV vaccine, and 2) provider recommendation of HPV vaccine for males and females in the recommended age range (11-12 years). The intervention toolkit will include evidence-based components aimed at the practice-level, provider-level and parent-level that will be tested through a cluster-randomized trial design. The primary hypothesis is that implementation of the comprehensive vaccine promotion toolkit in the pediatric health care setting will increase the likelihood that an adolescent receives initiates HPV vaccination.

At the initial visit, parents of adolescent patients at participating pediatric practices will complete a brief questionnaire assessing their knowledge, attitudes, and beliefs about adolescent health, including protection against infectious diseases during adolescence. The parents will be contacted again three months later to complete a short follow-up interview on the general health of their adolescent child, immunization status, and attitudes regarding vaccination.

DETAILED DESCRIPTION:
Since the introduction of HPV vaccine, there have been a number of studies examining attitudes and barriers related to HPV vaccine uptake among adolescent and young adult women, parents, and healthcare providers. Through these surveys, a number of distinct themes regarding reasons for not taking the HPV vaccine have emerged, including lack of provider recommendation, lack of awareness about the vaccine and the need for vaccination, concerns about vaccine effectiveness, concerns about vaccine safety, the potential of a vaccine against a sexually transmitted infection to increase promiscuity, cost of the vaccine doses, and the lack of routine adolescent well-care visits. However, many of these studies have used endpoints related to HPV vaccine knowledge or intention to vaccinate rather than actual vaccination uptake. Interventions that use endpoints related to vaccination uptake rather than knowledge or intention to vaccinate, as well as those that address multiple levels of the healthcare decision making process, will be crucial in addressing routine immunization coverage among adolescents. At the end of the evaluation of this intervention package, the researchers of this study hope to have identified a comprehensive and easily scalable "shelf-ready" toolkit aimed at increasing uptake of vaccines that are indicated during adolescence. If successful, this package could easily be implemented on a national level.

In the evaluation study, the researchers will use a cluster-randomized trial design to test whether exposure to the intervention package increases the likelihood of vaccine receipt by an adolescent in a practice randomized to receive the intervention package compared to an adolescent in a practice randomized to the control (standard of care) arm. Participating pediatric practices will be pair-matched based on overall adolescent patient load and historical HPV vaccine uptake and pairs will be randomized to one of two study arms:

1. Intervention arm: The pediatric practices randomized to this arm will receive the comprehensive adolescent vaccine promotion package. Practice physicians and staff will be familiarized with each component, and practices will be instructed to implement each vaccine-promotion component to the best of their ability.
2. Control arm: The pediatric practices randomized to the control arm will not receive the comprehensive vaccine promotion package and will instead be instructed to continue offering their standard adolescent vaccination promotion practices to adolescent patients.

Parents of eligible adolescents at participating practices will be given the opportunity to take part in this study. At the initial visit, parents of adolescent patients will complete a brief questionnaire assessing their knowledge, attitudes, and beliefs about adolescent health, including protection against infectious diseases during adolescence. The parents will be contacted again three months later to complete a short follow-up interview on the general health of their adolescent child, immunization status, and attitudes regarding vaccination.

ELIGIBILITY:
Parents are enrolled into the study based on their children meeting age and prior vaccination requirements.

Inclusion Criteria:

* Adolescent males and females aged 11-12 years and their parents
* No previous receipt of any HPV vaccine dose by the adolescent

Exclusion Criteria:

* Not English speaking (adolescents and parents)

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Initiation of HPV vaccine by adolescents | Month 3 Follow-Up
  During the follow-up interview, parents are asked if their child received the HPV vaccine during the visit with their pediatrician when they enrolled in this study. Possible responses are:
  * Yes, they received a dose of this vaccine
  * No, the received a dose of this vaccine before that visit
  * No, but they received a dose of this vaccine at a later visit
  * No, they have not received this vaccine
  * Don't know

SECONDARY OUTCOMES:
Vaccine Confidence Scale score | Month 3 Follow-Up
  Parental knowledge, attitudes, and beliefs about adolescent vaccination will be measured with the Vaccine Confidence Scale. The Vaccine Confidence Scale is an 8-item survey where respondents indicate the degree of their agreement with statements relating to vaccines (for example "Vaccines are safe"). Responses are on a scale of 0 to 10 where 0 = "Strongly Disagree", 5 = "Neutral", and 10 = "Strongly Agree". After reverse-coding certain items on the scale, the mean score of all responses serves as the total score. Total scores can range from 0 to 10 where higher scores indicate increased knowledge, attitudes, and beliefs regarding adolescent vaccination.
Provider perception of the intervention | At the end of the study (about 2 years)
  At the conclusion of the study period, the perceptions of healthcare providers and practice managers in the intervention practices regarding the intervention packages will be evaluated. Providers will respond to questions to share their perceptions on the extent to which the intervention was fully implemented (e.g., was querying of GRITS and the electronic medical record done consistently), and perceptions on the ease and helpfulness of the intervention components (e.g., talking points, printed materials) in facilitating conversations about HPV vaccination leading to vaccine receipt.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bednarczyk, PhD, Principal Investigator — Emory University
Locations (6):
- United States (6):
  - DV Pediatrics, Canton, Georgia
  - Crescent Pediatrics, Duluth, Georgia
  - Lawrenceville Pediatrics - Lawrenceville Office, Lawrenceville, Georgia
  - West Atlanta Pediatrics, Lithia Springs, Georgia
  - Lawrenceville Pediatrics - Loganville Office, Loganville, Georgia
  - Northlake Pediatric Associates, Stone Mountain, Georgia

IPD SHARING:
Plan to Share IPD: Undecided